CLINICAL TRIAL: NCT02866526
Title: Determinants and Consequences of the Transition to Adulthood Among Adolescents With Haemophilia - TRANSHEMO
Brief Title: Determinants and Consequences of the Transition to Adulthood Among Adolescents With Haemophilia
Acronym: TRANSHEMO
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-30
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Haemophilia
Keywords: adolescents; young adults
MeSH Terms: conditions — Hemophilia A | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: adolescents (14-17 years old)
  Interventions: Other: Patient questionnaire
- group 2: young adults (20-29 years old)
  Interventions: Other: Patient questionnaire

INTERVENTIONS:
Other: Patient questionnaire — quantitative and qualitative data collection will be proposed.

SUMMARY:
Severe haemophilia is a rare disease characterized by spontaneous bleedings from early childhood, which may lead to various complications especially in joints. Due to advances in medical care and more specifically in the development of prophylactic strategies by the application of clotting factor concentrates, life expectancy of persons with severe haemophilia has significantly increased over the last decades. This progress requires a long-term follow-up, including into adulthood. The adherence to a regular clinical follow-up and to a prophylactic treatment then depends on how successful patients' transition from childhood to adulthood has been as this process involves a transfer of responsibility from parents to patients concerning the management of their health. Beyond the issue of patients' adherence, a suboptimal transition may also impair quality of life and the entry into adulthood, especially at the social, emotional and professional levels. Only a few studies have been conducted to identify the specific needs and difficulties young persons with severe haemophilia experience during their transition from childhood to adulthood, and none of these studies has been carried out in France where the features of the health care system are very specific.

Therefore, this study aims to address the issue of transition into adulthood among young persons with severe haemophilia in France. This study will focus not only on the facilitators and barriers of the access to health care but also, from a more global perspective, on all the specific concerns and difficulties they may experience as they grow into adulthood which may impair their long-term health related quality of life as well as their personal empowerment. This study will also allow to identify some of the socio- cognitive, emotional, and familial determinants of a good transition into adulthood.

DETAILED DESCRIPTION:
The main objective of this study is to assess the impact of transition from adolescence into adulthood especially on adherence to health care, among young people with severe haemophilia in France.

The operational objectives of this study are: i) to compare the level of adherence in adolescents and in young adults (YA) ii) to identify determinants (medical, organisational, socio-demographic and social, and psychosocial and behavioural factors) of the level of adherence in YPWH (young people with haemophilia), iii) to assess specific factors involved in suboptimal level of adherence in the sub-groups of adolescents on one hand and of YA on the other hand, iv) to identify groups of patients (clusters) regarding both their level of adherence and their psychosocial characteristics, v) to examine trough a qualitative approach YPWH needs and expectations towards the health care system during the transition process, and to identify some ways to improve their global care.

This study is an exploratory, observational, multicentric, transversal study aimed at describing the perceptions of adolescents (14-17 years old) with severe haemophilia to those of young adults (20-29 years old) regarding their expectations and their feelings about growing into adulthood. Every patient enrolled in the FranceCoag national cohort (cohort of French patients suffering from inherited deficiencies of coagulation proteins), suffering from severe haemophilia, aged from 14 to 17 years old or from 20 to 29 years old, will be offered to get enrolled in the TRANSHEMO study (expected number eligible of participants: 154 adolescents and 389 young adults). , among whom 70% are expected to take part in the study). The patients' participation in this study will not modify their medical or paramedical care. A multifocal approach which combines both quantitative and qualitative data collection will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe haemophilia
* Patients enrolled in the FranceCoag national cohort
* Patients aged from 14 to 17 years old (adolescents group) or from 20 to 29 years old (young adults group)
* Adults patients having given their agreement to participate in the study, or minor patients authorized to participate in the study by their parents or their legal representatives

Exclusion Criteria:

* Patients with comprehension problems
* Patients unable to read or to write
* Adults patients not having given their agreement to participate in the study, or minor patients unauthorized to participate in the study by their parents or their legal representatives

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: cohort of persons with severe haemophilia
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Number of follow-up visits / theoretical number of follow-up visits over the last two years | Two years
  Adherence to clinical follow-up
Number of injections of prophylactic treatment realized / theoretical number of injections of prophylactic treatment over the last three months | 3 months
  Adherence to prophylactic treatment

SECONDARY OUTCOMES:
Patient-reported adherence | one day
  Specific item of the patient questionnaire (0-10 points)
Physician-reported adherence of the patient | one day
  Specific item of the medical questionnaire (0-10 points)
Number of haemorrhagic events | one day
  Specific item of the medical questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — ASSISTANCE Publique Hôpitaux de Marseille
Locations (28):
- France (28):
  - CHU D'Amiens, Amiens
  - CHU de Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - Chu Brest, Brest
  - CHU CAEN, Caen
  - Ch Chambery, Chambéry
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CH Versailles/ Le Chesnay, Le Chesnay
  - Chu Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civiles de Lyon, Lyon
  - Assistance Publique Hôpitaux de Marseille Hôpital de la Timone, Marseille
  - CH Montmorency, Montmorency
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Assistance Publique Hôpitaux de Paris, Paris
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Chu Rouen, Rouen
  - CHU Réunion, Saint-Denis
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Derived] Resseguier N, Rosso-Delsemme N, Beltran Anzola A, Baumstarck K, Milien V, Ardillon L, Bayart S, Berger C, Bertrand MA, Biron-Andreani C, Borel-Derlon A, Castet S, Chamouni P, Claeyssens Donadel S, De Raucourt E, Desprez D, Falaise C, Frotscher B, Gay V, Goudemand J, Gruel Y, Guillet B, Harroche A, Hassoun A, Huguenin Y, Lambert T, Lebreton A, Lienhart A, Martin M, Meunier S, Monpoux F, Mourey G, Negrier C, Nguyen P, Nyombe P, Oudot C, Pan-Petesch B, Polack B, Rafowicz A, Rauch A, Rivaud D, Schneider P, Spiegel A, Stoven C, Tardy B, Trossaert M, Valentin JB, Vanderbecken S, Volot F, Voyer-Ebrard A, Wibaut B, Leroy T, Sannie T, Chambost H, Auquier P. Determinants of adherence and consequences of the transition from adolescence to adulthood among young people with severe haemophilia (TRANSHEMO): study protocol for a multicentric French national observational cross-sectional study. BMJ Open. 2018 Jul 25;8(7):e022409. doi: 10.1136/bmjopen-2018-022409. PMID 30049701